CLINICAL TRIAL: NCT05971030
Title: Clinical Exploratory Research of Medial Prefrontal Cortex Combined With Dorsolateral Prefrontal Cortex Electrical Stimulation in the Treatment of Alzheimer's Disease
Acronym: CBS-m/dlPFC-AD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023062
Record Dates: First submitted 2023-07-20; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease; Electric Stimulation Therapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBS for mPFC and dlPFC (Experimental): Case series of AD patients who accept CBS for mPFC and dlPFC
  Interventions: Device: Cortical brain stimulation of mPFC and dlPFC

INTERVENTIONS:
Device: Cortical brain stimulation of mPFC and dlPFC — Left medial prefrontal cortex combined with dorsolateral prefrontal cortex electrical stimulation

SUMMARY:
Alzheimer's disease (AD) is a common neurodegenerative disease characterized by progressive cognitive impairment and memory impairment, and is also a major cause of global dementia, characterized by progressive decline in memory and daily living behavior. The incidence rate of AD increases with age. The prevalence rate of AD among men over 65 years old in China is 3.4%, and that of women is 7.7%, with a total prevalence rate of 5.9%. Among them, people over 65 years old can live for an average of 4 to 8 years after being diagnosed with Alzheimer's disease. According to statistics, there were approximately 5.98 million AD patients in China in 2005, reaching 10.2 million in 2020 and 22.5 million by 2040, making it the largest country with AD.

At present, the treatment of AD is mostly limited to drug therapy, including Acetylcholine enzyme inhibitor, N-methyl-D-aspartate receptor antagonist and brain cell metabolism promoter. Although there are many types of drugs, their efficacy is not satisfactory, as they not only cannot effectively prevent and cure AD, but also cannot slow down the progression of AD. Regarding the surgical treatment of AD, neuromodulatory surgery, especially DBS (Deep Brain Electrical Stimulation), involves implanting stimulation electrodes into deep neural nuclei in the brain and performing electrical stimulation to change the excitability of the corresponding nuclei or neural circuits, and has been included in alternative treatment plans. In the past 20 years, DBS technology has been continuously explored for the treatment of AD, but an increasing number of clinical trials have shown that there is no effective target for AD-DBS. Therefore, there is an urgent need for new treatment methods to improve the current treatment status.

DETAILED DESCRIPTION:
The main principle of DBS is to regulate the activity of neural components by implanting electrodes into key brain regions using a built-in pulse generator. The basic principle of using DBS in AD is that AD is not only a neurodegenerative disease, but also a neural circuit disease, because it affects several integrated cortical and subcortical pathways, especially those involving memory and cognition. DBS implants stimulation electrodes into deep neural nuclei in the brain for electrical stimulation, altering the excitability of the corresponding nuclei or neural circuits, which may lead to therapeutic effects. However, the stimulation targets of the electrodes are still unclear.

There are currently 3 clinical studies on AD-DBS reported in the literature, using stimulation targets such as the Basal Nucleus of Meynert (NBM) and the fornix. One of the studies was reported this year by a team from Kuhn et al. in Germany. They used NBM as a stimulation target and treated 6 patients with DBS. The stimulation lasted for 12 months and was evaluated using the Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS Co g) and the Simplified Mental State Examination Scale (MMSE). Among them, one patient showed improvement in their ADAS Log score, two patients stabilized, and three patients continued to deteriorate in cognitive function. The other was a phase I clinical trial conducted by the Lozano team in Canada in 2010. The team used the fornix as a stimulation target to perform DBS treatment on 6 mild AD patients, with the same stimulation for 12 months. The results showed that only 1 out of 6 patients had significant improvement in cognitive function (reduced ADAS Cog score), while the remaining 5 patients still showed varying degrees of deterioration. In addition, Fontaine et al. reported in 2013 on a patient with transfornix electrical stimulation, where 12 months of continuous electrical stimulation stabilized the patient's MMSE and ADAS-Log scores. However, the above three studies all found that DBS can improve the glucose metabolism level of brain tissues in temporal and parietal lobes. The above studies indicate that although NBM and fornix electrical stimulation have some improvement in cognitive function in some AD patients, the overall improvement rate is low, with most patients in an unresponsive state. Therefore, given the core position of stimulation targets in deep brain electrical stimulation surgery, it is urgent to explore new stimulation targets in order to improve the efficacy of DBS. The combination of medial prefrontal cortex (mPFC) and dorsolateral prefrontal cortex (dlPFC) can serve as an ideal stimulation target At present, the treatment of AD is still a global challenge, but the non-invasive neural regulation techniques (rTMS and tDCS) based on the medial prefrontal cortex (mPFC) and dorsolateral prefrontal cortex (dlPFC) have preliminarily confirmed that mPFC and dlPFC regions may be potential therapeutic targets for AD, which can significantly improve the cognitive status of therapists. At present, the targets used for treating AD with DBS are the fornix and NBM, but the effectiveness of treating AD has not been confirmed. Based on a thorough analysis of current international research and in conjunction with previous research conducted by our center, the investigators propose to combine the left mPFC and dlPFC regions as stimulation targets and innovatively use sheet electrodes for cortical brain stimulation (CBS), which is well established. As a stimulation method of DBS, CBS stimulates the cortex relative to the deep stimulation target. For example, common pain electrical stimulation uses CBS, so the cortical electrical stimulation in this study adopts the naming method of CBS. On this basis, the investigators strictly set inclusion and exclusion criteria to ensure the quality of enrolled patients, and conducted thorough experimental design and validated the efficacy of CBS in treating AD from multiple perspectives using specific memory and cognitive function assessment scales, fusion function, structure, metabolic brain networks, and other methods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 40 to 70;
2. eets the diagnostic criteria for mild to moderate AD;
3. A CDR score of 0.5 or 1.0;
4. The MMSE score is between 18 and 28;
5. Regularly taking cholinesterase inhibitors for more than 6 months

Exclusion Criteria:

1. Existence of brain structural abnormalities (such as brain tumors, cerebral infarction, and intracranial hematoma);
2. Suffering from other neurological or psychiatric diseases;
3. Accompanying comorbidities that are not suitable for surgical treatment;
4. Individuals with contraindications for MRI or PET testing

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Auditory verbal learning test (AVLT) before and after DBS | 1 months before DBS, 1 month, 2 months, 3 months, 6 months, and 12 months after DBS.
  ALVT will be performed before and after DBS operations to examine the AD. patients' ability.

SECONDARY OUTCOMES:
Mini-mental State Examination (MMSE) before and after DBS | 1 months before DBS, 1 month, 2 months, 3 months, 6 months, and 12 months after DBS.
  MMSE will be performed before and after DBS operations to examine the AD.
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 1 months before DBS, 1 month, 2 months, 3 months, 6 months, and 12 months after DBS.
  ADAS-COG will be performed before and after DBS operations to examine the AD.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
We will publish our results once the study finished
Supporting Information: CSR
Time Frame: after the study finished